CLINICAL TRIAL: NCT03733665
Title: HES and NICOR Data Linkage for Cardiac Failure Population Analysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: DARS-NIC-174209-R8G8N-v0
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure; Registries; Patient Readmission
Keywords: Hospital Episode Statistics; HES; National Institute for Cardiovascular Outcomes Research; NICOR; National Heart Failure Audit
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart failure patients: All patients in NICOR's National Heart Failure Audit will be matched to those in NHS Digital's HES database who have a 4-character primary diagnosis of I50.0-I50.9.
  Interventions: Other: Patients admitted to hospital

INTERVENTIONS:
Other: Patients admitted to hospital — Data is captured in HES for all patient interactions with the NHS (each episode) in England. All patients admitted for heart failure have data captured in the National Heart Failure Audit.

SUMMARY:
This study is a population-based, patient-level analysis of heart failure in England over a 5-year period using a dataset created by linking HES and NICOR databases. Our analyses will look into the re-occurrence of hospitalisation after the initial diagnosis of heart failure, the influence of population factors on risk of re-hospitalisation, and the resultant cost implications in an NHS environment.

DETAILED DESCRIPTION:
Data from the National Heart Failure Audit (NICOR) and Hospital Episodes Statistics (NHS Digital) will be linked, by NHS Digital, using fields that are recorded in both databases (for example, NHS number). We will receive de-anonymised data that has been pseudo-anonymised, allowing for patient-level analyses but without identifying individual patients.

ELIGIBILITY:
Inclusion Criteria:

* patients >17 years old
* individual patient data appears on both HES and NICOR databases
* 4-character primary diagnosis codes I50.0-I50.9

Exclusion Criteria:

* patient requests withdrawal from analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute decompensated heart failure (ADHF) is a sudden worsening of the signs and symptoms of heart failure, which typically includes difficulty breathing (dyspnoea) and leg oedema. ADHF is a common and potentially serious cause of acute respiratory distress. Treatment of ADHF consists of reducing the excess fluid retention with diuretics along with improving heart function with pharmacological treatment. Although pharmacological treatments exist for heart failure patients with reduced ejection fraction (ACE inhibitors, beta-blockers), a substantial fraction of patients exhibit preserved ejection fraction where treatment consists solely of management of comorbidities and symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Readmission | 2012-2017
  Any repeat hospitalisation for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Chalkidou, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Privacy notice and patient notification information — http://www.kitec.co.uk/perch/resources/nicor-patient-notification-text.docx